CLINICAL TRIAL: NCT03104998
Title: Neotililty Trial: Effect of Coenzyme Q10 on Semen Parameters in Men With Idiopathic Infertility
Acronym: Neotility
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No further patient enrollment
Sponsor: PharmEvo Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PE/PK/Neotility/SP/2017-01
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2017-03

CONDITIONS: Idiopathic Infertility
Keywords: Idiopathic; Infertility; coenzyme q10; Pakistan
MeSH Terms: conditions — Infertility | interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- coenzyme Q10 (Other): Dose of 200 mg of CoQ10 taken daily by mouth from day 1 till 26 weeks
  Interventions: Drug: Coenzyme Q10

INTERVENTIONS:
Drug: Coenzyme Q10 — 200 mg of CoQ10 or placebo daily by mouth from day 1 till 26 weeks. CoQ10 treatment is safe, even at the highest doses cited in the literature. Most clinical trials have not reported significant adverse effects that necessitated stopping therapy. However, gastrointestinal effects such as abdominal discomfort, nausea, vomiting, diarrhea, and anorexia have occurred. Allergic rash and headache have also been reported
  Other Names: NeoQ10

SUMMARY:
To study the effect of coenzyme Q10 on semen parameters in men with idiopathic infertility

DETAILED DESCRIPTION:
Decreased serum CoQ10 concentrations as well as a decrease in the CoQ10H2 to-ubiquinone ratio have been demonstrated in diseases associated with OS. A strong correlation among sperm count, motility and ubiquinol-10 levels in seminal fluid has also been reported.

The aim of the present study is to investigate whether the effects of the exogenous administration of ubiquinol in the improvement of semen parameters in Pakistani men population.

Patients who full filled the inclusion criteria and gave informed written consent will be included in the trial. Patient will start to take medication and will take it for 26 weeks.

All men undergo a thorough physical examination, a detail history, serum biochemical and hematological laboratory tests and measurement of serum sex and thyroid hormone levels. A questionnaire will be used to collect information on demographic characteristics. Two semen samples 1 and 2 month apart will be obtained after 3 to 5 days of sexual abstinence and process within 1 hour of ejaculation. The mean of the two will be used for statistical analysis. Semen analyses will be performed using WHO recommended methods.

3 ml of blood will be withdrawn from the patient for the serum hormones analysis and total amount of semen will required for analysis of semen parameters.

Sponsor will bear the test cost of patient during the study treatment period.

ELIGIBILITY:
Inclusion Criteria:

* To sign the Informed Consent form
* Patients will be recruited in the study if they will fulfilled the criteria of history of primary infertility of more than 2 years, abnormal sperm count and motility
* age between 20 and 50 years
* No known medical or surgical condition which can result in infertility

Exclusion Criteria:

* Voluntary withdrawal
* Poor compliance of visit/treatment
* A history of cancer chemotherapy or radiotherapy
* A history of genital disease such as cryptorchidism and varicocele; a history of genital surgery
* Body mass index 30 kg/m or greater; any endocrinopathy
* Ychromosome microdeletions or karyotype abnormalities
* leukocytospermia
* Drug or substance abuse; tobacco use;
* Use of anticonvulsants, androgens or antiandrogens
* Significant liver (serum bilirubin greater than 2.0 mg/dl)
* Renal function (serum creatinine greater than 2.0 mg/dl) impairment
* Patients with severe oligozoospermia (less than 5 X 106/ml), azoospermia and testicular volume less than 12 ml will also excluded from study.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Measure the change in semen parameters after 26 Weeks of coenzyme q10. | 26 weeks
  To measure the change in semen parameters after 26 Weeks of coenzyme q10.
  Designated as safety issue: No

SECONDARY OUTCOMES:
Adverse Event | 26 weeks
  Proportion of participants experiencing an adverse event (AE) leading to permanent discontinuation of study medication [Designated as safety issue: Yes]

CONTACTS AND LOCATIONS:
Overall Officials: Masood Jawaid, MRCS,FCPS, Study Chair — PharmEvo Pvt Ltd
Locations (1):
- HillPark Hospital, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Ligny W, Smits RM, Mackenzie-Proctor R, Jordan V, Fleischer K, de Bruin JP, Showell MG. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2022 May 4;5(5):CD007411. doi: 10.1002/14651858.CD007411.pub5. PMID 35506389